CLINICAL TRIAL: NCT01799564
Title: A Phase I Study to Establish the Safety and Efficacy of Retinal Pigment Epithelium Micropulse Laser in Subjects With Geographic Atrophy Secondary to Dry Age-related Macular Degeneration
Brief Title: Micropulse Laser for Geographic Atrophy
Acronym: MPL4DRY
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Institut de la Macula y la Retina (Other)
Responsible Party: Principal Investigator, Jordi Mones MD PhD, MD, PhD, Institut de la Macula y la Retina
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: MPL4DRY
Record Dates: First submitted 2013-02-25; First posted 2013-02-27 (Estimated); Last update posted 2019-09-18 (Actual); Status verified 2019-09

CONDITIONS: Geographic Atrophy; Age-related Macular Degeneration
Keywords: Geographic atrophy; Age-related macular degeneration; Fundus autofluorescence
MeSH Terms: conditions — Geographic Atrophy; Macular Degeneration

STUDY DESIGN:
Who Masked: Care Provider, Outcomes Assessor
Oversight: Data Monitoring Committee: No

ARMS (2):
- Micropulse (Experimental): Micropulse laser will be applied to the inferior hemiretina next to the area of atrophy in a randomly selected eye in 1, 2 or 3 occasions
  Interventions: Procedure: Micropulse
- Control (No Intervention): The fellow eye does not receive any treatment

INTERVENTIONS:
Procedure: Micropulse — Between 1 and 3 sessions of micropulse laser will be applied in the inferior hemiretina of the randomly selected eye
  Arms: Micropulse

SUMMARY:
Geographic atrophy (GA) causes the loss of the retinal pigment epithelium (RPE) cells in broad areas of the retina. The application of subthreshold micropulse laser spots in healthy RPE in the vicinity of the area of GA may restore the imbalance in survival factors caused by the disease (ie, the laser may decrease vascular endothelial growth factor and RPE-derived transforming growth factor beta, upregulation of pigment epithelium-derived factor). This may slow or even stop the enlargement of atrophy secondary to GA, and therefore, avoid further vision loss.

ELIGIBILITY:
Inclusion Criteria:

* GA > 0.5 disk areas secondary to AMD in both eyes
* 50 years or older
* The periphery of the atrophic lesions must demonstrate increased autofluorescence
* Best corrected visual acuity between 20/20 and 20/400 inclusive
* Clear ocular media
* Ability to provide informed consent and attend all study visits

Exclusion Criteria:

* GA secondary to other causes aside from AMD
* Evidence of choroidal neovascularization in either eye
* Any prior treatment for AMD, aside from antioxidants
* Any other ocular condition that would progress in the study period and confound visual acuity assessment
* Any ocular or systemic medication known to be toxic to the lens, retina or optic nerve
* Presence of idiopathic or autoimmune-associated uveitis
* Any intraocular surgery 3 months of entry
* Any prior thermal laser in the macula
* History of vitrectomy, filtering surgery, corneal transplant or retinal detachment surgery
* Previous therapeutic radiation in the ocular region in either eye
* Any treatment with an investigational agent in the previous 60 days before study entry

Min Age: 50 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 11 (Actual)
Dates: Start 2012-08; Primary Completion 2013-11-27 (Actual); Study Completion 2013-11-27 (Actual)

PRIMARY OUTCOMES:
Change in area of atrophy as measured with fundus autofluorescence (FAF) | Change in area from baseline to week 48
  Difference in baseline area of atrophy as measured with FAF at week 48

CONTACTS AND LOCATIONS:
Overall Officials: Jordi Monés, MD, PhD, Principal Investigator — Institut de la màcula i de la retina
Locations (1):
- Institut de la màcula i de la retina, Barcelona, Spain